CLINICAL TRIAL: NCT03173313
Title: COOL-AMI EU Pivotal Trial: A Multicenter, Prospective, Randomized-Controlled Trial to Assess the Safety and Effectiveness of Cooling As an Adjunctive Therapy to Percutaneous Intervention in Patients With Acute Myocardial Infarction
Brief Title: COOL AMI EU Pivotal Trial to Assess Cooling as an Adjunctive Therapy to PCI In Patients With Acute MI (Phase A)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZOLL Circulation, Inc., USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EDC-3135
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Results first posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-01

CONDITIONS: Acute Myocardial Infarction
Keywords: Hypothermia; Acute Myocardial Infarction; AMI; PCI; Therapeutic Hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cooling + PCI (Other): The subjects will be considered to be enrolled in the Test Arm of the trial when all inclusion and exclusion criteria have been met, the informed consent form has been signed, and randomization to the Test Arm of the trial to allow cooling with the Proteus IVTM System before and after PCI.
  Interventions: Device: Intravascular permissive hypothermia as an adjunct to PCI
- PCI only (Other): The subjects will be considered to be enrolled in the Control Arm of the trial when all inclusion and exclusion criteria have been met, the informed consent form has been signed, and randomization to the Control Arm of the trial to allow PCI only.
  Interventions: Device: Intravascular permissive hypothermia as an adjunct to PCI

INTERVENTIONS:
Device: Intravascular permissive hypothermia as an adjunct to PCI — Cooling with ZOLL Proteus IVTM System before and after Percutaneous Coronary Intervention (PCI) -or- Standard of Care for PCI

SUMMARY:
The objective of this trial is to evaluate the safety and effectiveness of therapeutic hypothermia, using the ZOLL Proteus IVTM System, as an adjunctive therapy for patients presenting with acute anterior myocardial infarction (AMI) and undergoing percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
A multicenter, prospective, interventional, randomized-controlled trial. Randomization will be in a 1:1 ratio, Test Arm (PCI + Cooling) or Control Arm (PCI alone) in up to 468 randomized subjects (234 subjects in each arm). Endpoint: Relative reduction of 20% in mean anterior myocardial infarct size as determined by Cardiac Magnetic Resonance (cMR) imaging at 4-6 days post infarct in the Test Arm (cooling + PCI) relative to the Control Arm (PCI only).

ELIGIBILITY:
Inclusion Criteria:

1. The patient is ≥ 18 years of age.
2. The patient must have symptoms consistent with AMI (i.e. chest pain, arm pain, etc.) and unresponsive to nitroglycerin, with symptoms beginning greater than 30 minutes but less than 6 hours prior to presentation at hospital.
3. Qualifying Infarct location:

   1. Roll-In subjects: Evidence of Acute Anterior or Inferior MI with ST-segment elevation of >= 0.2 mV in two or more anterior or inferior contiguous precordial leads.
   2. Randomized subjects: Evidence of Acute Anterior MI only with ST-segment elevation of >= 0.2 mV in two or more anterior contiguous precordial leads.
4. The patient is eligible for PCI.
5. The patient is willing to provide written informed consent to participate in this clinical trial.

Exclusion Criteria:

1. The patient has had a previous Myocardial Infarction.
2. The patient is experiencing cardiogenic shock (systolic blood pressure [SBP] <80 mmHg and non-responsive to fluids, or SBP <100 mmHg with vasopressors, or requirement for an intra-aortic balloon pump [IABP]).
3. The patient is presenting with resuscitated cardiac arrest, atrial fibrillation, or Killip risk stratification class II through IV.
4. The patient has an aortic dissection or requires an immediate surgical or procedural intervention other than PCI.
5. The patient has known history of Congestive Heart Failure (CHF), hepatic failure, end-stage kidney disease or severe renal failure (clearance < 30ml/min/1.73m²).
6. The patient is febrile (temperature > 37.5 °C) or has experienced an infection with fever in the last 5 days.
7. The patient has a known previous CABG.
8. The patient has a known recent stroke within 90 days of admission.
9. Cardio-pulmonary decompensation that has occurred en route to the hospital or, in the opinion of the physician, that is imminent or likely to occur following presentation to the clinical site.
10. Contraindications to hypothermia, such as patients with known hematologic dyscrasias which affect thrombosis (e.g., cryoglobulinemia, sickle cell disease, serum cold agglutinins) or vasospastic disorders (such as Raynaud's or thromboangitis obliterans).The patient has a known hypersensitivity or contraindication to aspirin, heparin, or sensitivity to contrast media, which cannot be adequately pre-medicated.
11. Any contraindication to cardiac MRI, or any implant in the upper body which may cause artifacts on cardiac MRI imaging.
12. The patient has a known hypersensitivity or contraindication to aspirin, heparin, or sensitivity to contrast media, which cannot be adequately pre-medicated.
13. The patient has a known history of bleeding diathesis, coagulopathy, cryoglobulinemia, sickle cell anemia, or will refuse blood transfusions.
14. The patient has a height of <1.5 meters (4 feet 11 inches).
15. The patient has a known hypersensitivity or contraindication to buspirone hydrochloride or Pethidine (Meperidine) and/or has been treated with a monoamine oxidase inhibitor in the past 14 days.
16. Patient has a known history of severe hepatic or renal impairment, untreated hypothyroidism, Addison's disease, benign prostatic hypertrophy, or urethral stricture that in the opinion of the physician would be incompatible with Pethidine administration.
17. The patient has an Inferior Vena Cava filter in place (IVC).
18. The patient has a pre-MI life expectancy of <1 year due to underlying medical conditions or pre-existing co-morbidities.
19. The patient has a known, unresolved history of drug use or alcohol dependency, or lacks the ability to comprehend or follow instructions.
20. The patient is currently enrolled in another investigational drug or device trial.
21. The patient is apprehensive about or unwilling to undergo the required MRI imaging at follow-up, has a documented or suspected diagnosis of claustrophobia, or has Gadolinium allergy, or is in permanent Atrial Fibrillation.
22. The patient has received thrombolytic therapy en route to the hospital.
23. The patient shows clinical evidence of spontaneous reperfusion as observed symptomatically and/ or from ECG findings (partial or complete ST resolution in ECG prior to informed consent and randomization).
24. The patient is a vulnerable subject, for instance, a person in detention (i.e., prisoner or ward of the state).
25. The patient is a female who is known to be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2019-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marko Noc, Principal Investigator — University Medical Center Ljubljana Slovenia
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cooling + PCI | PCI Only
Started | 58 | 53
Informed Consent Signed | 58 | 53
Randomized | 58 | 53
Cooled | 54 | 0
4-6 Day Follow-up | 57 | 53
30-day Follow-up | 52 | 51
12-month Follow-up | 49 | 48
Completed | 49 | 48
Not Completed | 9 | 5
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Death | 5 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Diagnosis of Takotsubo Cardiomyopathy | 0 | 1
Not completed — Bone Fracture | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cooling + PCI | PCI Only | Total
Number analyzed (Participants) | 58 | 53 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 31 | 72
  >=65 years | 17 | 22 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (10.7) | 61.0 (11.0) | 59.6 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 43 | 39 | 82
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 57 | 52 | 109
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Bosnia and Herzegovina | 5 | 4 | 9
  Estonia | 11 | 11 | 22
  Hungary | 17 | 15 | 32
  Serbia | 19 | 16 | 35
  Slovakia | 5 | 4 | 9
  Slovenia | 0 | 1 | 1
  United Kingdom | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Relative Reduction of 20% in Mean Anterior Myocardial Infarct Size as Determined by Cardiac Magnetic Resonance (cMR) Imaging at 4-6 Days Post Infarct in the Test Arm (Cooling + PCI) Relative to the Control Arm (PCI Only).
Description: The primary outcome is to compare the mean infarct size in the Test Arm (cooling + PCI) to the mean infarct size in the Control Arm (PCI only) at 4-6 days post infarct.
Time Frame: 4-6 Days
Population: Per-protocol population with available infarct size. 19 Test Arm subjects were excluded from the analysis due to not meeting eligibility criteria, having a repeat MI before 4-6 day cMRI, unavailable cMRI, or did not follow cooling per protocol.
  9 Control Arm subjects were excluded from the analysis population due to not meeting eligibility criteria, having a repeat MI before 4-6 day cMRI, or unavailable cMRI.
Measure: Mean (Standard Deviation); unit: LV%
Arm/Group | Cooling + PCI | PCI Only
Number analyzed (Participants) | 39 | 44
LV% | 21.6 (11.5) | 20.9 (12.6)

2. Primary Outcome: Per-patient Rate of Composite Major Adverse Cardiac Events (MACE) in Randomized Subjects
Description: The primary safety outcome is to compare the per-patient rate of composite Major Adverse Cardiac Events (MACE) in the Test Arm (cooling + PCI) to the Control Arm (PCI only) at 30-Day follow-up to determine non-inferiority to the Control. Composite MACE is defined as Cardiac Death (CD), All Myocardial Re-Infarction (All MI) and Clinically-Indicated Target Vessel Revascularization (CI-TVR).
Time Frame: 30 Days
Population: Per-protocol population. 16 Test Arm subjects were excluded from the analysis due to not meeting eligibility criteria, having a repeat MI before 4-6 day cMRI, or did not follow cooling per protocol.
  4 Control Arm subjects were excluded from the analysis population due to not meeting eligibility criteria or having a repeat MI before 4-6 day cMRI.
Measure: Count of Participants; unit: Participants
Arm/Group | Cooling + PCI | PCI Only
Number analyzed (Participants) | 42 | 49
Participants
  Cardiac Death | 1 | 0
  Cardiac Death and Myocardial re-infarction and clinically-indicated target vessel revascularization | 1 | 0
  No MACE Event | 40 | 49

ADVERSE EVENTS:
Time Frame: 30 Days
Description: Adverse Events
Arm/Group | Cooling + PCI | PCI Only
All-Cause Mortality (participants affected / at risk) | 5/58 | 0/53
Serious Adverse Events (participants affected / at risk) | 18/58 | 4/53
Other Adverse Events (participants affected / at risk) | 45/58 | 22/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cooling + PCI (N=58) | PCI Only (N=53)
Cardiac arrest (Cardiac disorders) | 2 | 0
Cardiogenic shock (Vascular disorders) | 6 | 0
Infections - listed (Infections and infestations) | 5 | 0 — Pneumonia, Sepsis, Upper respiratory tract infection
Myocardial infarction (Musculoskeletal and connective tissue disorders) | 1 | 0
Other cardiac - listed (Cardiac disorders) | 5 | 1
Pulmonary edema (Cardiac disorders) | 1 | 0
Respiratory failure (Metabolism and nutrition disorders) | 2 | 0
Stent thrombosis (Vascular disorders) | 2 | 1
Ventricular fibrillation (Cardiac disorders) | 6 | 2
Ventricular tachycardia (Cardiac disorders) | 2 | 0
Acute renal insufficiency (Renal and urinary disorders) | 1 | 0
Bleeding (Vascular disorders) | 2 | 0
Hematoma (Vascular disorders) | 1 | 0
Hypernatraemia/Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Vascular perforation or dissection (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cooling + PCI (N=58) | PCI Only (N=53)
Atrial fibrillation (Cardiac disorders) | 25 | 2
Infections - listed (Infections and infestations) | 7 | 0 — Pericarditis, Pneumonia, Urinary tract infection
Other cardiac - listed (Cardiac disorders) | 16 | 11 — Cardiomyopathy, Chest pain, Congestive heart failure, Hypertension, Hypotension, Intracardiac thrombus, Left Main embolization
Uncontrolled shivering (Musculoskeletal and connective tissue disorders) | 12 | 0
Ventricular tachycardia (Cardiac disorders) | 3 | 1
Anxiety (Psychiatric disorders) | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 7 | 3
Sleep disorder (Psychiatric disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 3 | 0

LIMITATIONS AND CAVEATS:
The COOL-AMI EU Pivotal Trial enrolled a total of 111 subjects. The study was terminated prematurely after non-cooling related factors were identified as having a significant impact on group differences, including significantly higher total ischemic time and door-to-balloon time in the cooling arm. This early stoppage limits the power of the results to detect a difference between the treatment arms. Further study needs to be done to evaluate the effectiveness of therapeutic hypothermia in STEMI.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/13/NCT03173313/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/13/NCT03173313/SAP_001.pdf